CLINICAL TRIAL: NCT02809547
Title: Remote Arthritis Disease Activity MonitoR (RADAR 1) - a Feasibility Study of Home-based Dried Blood Spot Use to Monitor an Inflammatory Marker in Rheumatoid Arthritis Patients.
Brief Title: RADAR1- Trial of a New Blood Sample Method (Remote Arthritis Disease Activity MonitoR)
Acronym: RADAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 16/0019
Record Dates: First submitted 2016-06-17; First posted 2016-06-22 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

ARMS (2):
- In Clinic monitoring (Active Comparator): 70 method comparison patients who represent a C-reactive protein (CRP) reference range and have retrievable study outcome measures will have a whole blood sample and DBSS taken at recruitment and at a routine six week review.
  Interventions: Device: Dried Blood Spot device
- At Home monitoring (Experimental): 30 Prospective patients will provide (i) one whole blood sample and one set of dried blood spot samples (DBSS) at recruitment, (ii) a set of DBSS once a week for six weeks from recruitment, with a matched whole blood sample at six week appointment, (iii) two extra sets of DBSS to be taken during a flare and 24 hours after (iv) 6 prospective patients will have daily hand movement data collected for 5 minutes on each occasion using a provided data glove.
  Interventions: Device: Dried Blood Spot device

INTERVENTIONS:
Device: Dried Blood Spot device

SUMMARY:
It is important that patients who suffer from Rheumatoid Arthritis (RA) have their disease monitored at an early stage, as well as when it is established. Presently, if a patient is to be assessed by means of disease activity scores and blood tests, they must attend a hospital appointment, which can be difficult for patients who live far from the clinic. It would be beneficial to be able to monitor and reliably define and report a disease 'flare' at home. Quite often, by the time the patient attends for an appointment, flare ups have subsided. This study will evaluate the possibility for patients to take their own blood samples in the comfort of their own home, by transferring finger prick blood droplets to a dried blood spot sample (DBSS) card. Patients would then send the cards to the laboratory to test for clinically relevant protein markers. The feasibility of 'remote' monitoring of the patient's disease will be explored.

DETAILED DESCRIPTION:
In an arthritis patient population living some distance from hospitals, collection of a series of blood samples to monitor disease activity in a timely fashion is difficult. The ability to monitor markers of inflammation, such as C-reactive protein (CRP) and gauge a patient's response to treatments via disease activity score (i.e. DAS28-ESR) is not just important in early stage disease but also in patients with established disease. Patients with chronic disease tend to lose self-confidence in managing their condition and a substantial proportion can suffer recurrent disease flare- ups. These flare-ups are costly in terms of appointments with GP and specialist clinics and result in significant work disability.

Being able to reliably define and report a disease 'flare' in arthritis is currently problematic as there are no objective measures available to the patient while at home. The clear definition of a flare, as determined through blood testing would help justify an increase in immunosuppressant dose or a course of steroids. Currently, patients make a visit to their GP or hospital clinic, at 6 week intervals at best. In reality, this means that opportunities to monitor CRP during an active 'flare' are often missed and an informed intervention (medication adjustments) is not possible. Home monitoring is constrained by the costs of making phlebotomists available to make frequent home visits to patients. Also for markers which are unstable at ambient temperatures, blood samples need to be refrigerated and rapidly transported to the laboratory for analysis.

Thus the ability for the patient to collect their own blood samples in their own home and send these at ambient temperature to a laboratory would enable 'remote' and timely monitoring of chronic disease. The investigators have recently completed an Arthritis Research UK funded clinical study that demonstrated that a number of clinically relevant proteins related to flares (i.e.?) were reliably collected, stored for less than three months and extracted from dried blood spots (n=20 arthritis patients). The paper cards used to collect blood droplets were pre-treated to stabilise proteins and minimise haemolysis contamination (caused by bursting and breakdown of red blood cells). Our results across 20 arthritis patients revealed that 90% recovery rates can be achieved from dried blood spot sample (DBSS) stored at room temperature for 3 month (relative to a matched -20'C frozen plasma sample). The inflammation marker proteins included C-reactive protein (CRP), tumour necrosis factor alpha and Immunoglobulin G. Without pre-treatment of the DBSS paper, only 53% of these proteins are recovered.

For the patient, use of DBSS means that GP and hospital visits to take blood and carry out tests could be reduced. With minimal training, samples would be obtained simply at home by the patient, over a six week period and then transported at room temperature using conventional post. Proteins could then be analysed at a central lab. In the future, the technology could accompany patient assessments of disease activity and complement ongoing studies focused on wearable sensors to measure joint movement and stiffness (UU Data-glove project).

For the hospital trust, use of this novel technology could obviate the need for patients to attend the clinic for blood sampling. Soon after prescribing a new treatment, clinicians could use DBSS to monitor treatment efficacy in reducing inflammation. This technology therefore offers an earlier opportunity than currently available to titre dosage and switch from ineffective drugs or treatments associated with adverse events. Furthermore, feedback of the monitoring information provided by DBSS could be given to the patient, via for example smartphone application, and has the potential to improve adherence to treatment plans.

ELIGIBILITY:
Inclusion Criteria:

Rheumatoid Arthritis will be diagnosed according to the joint American College of Rheumatology (ACR) and European League against Rheumatism (EULAR) 2010 criteria. Patients who are about to receive their first / a change in combination or dose of DMARD (prospective) or are currently being treated by DMARD therapy will be included in the study.

Exclusion Criteria:

Patients who have received or are receiving biologic therapy will be excluded from the study. Patients will be representative of the 'real life' patient population in the clinics who meet these criteria, and will not be excluded for other general health reasons.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-11; Primary Completion 2017-06 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
C-Reactive Protein concentrations | Baseline and Six week samples

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Ireland Centre for Stratified Medicine/ Altnagelvin Hopsital, Londonderry, United Kingdom

REFERENCES:
- [Derived] D'Cruz LG, McEleney KG, Cochrane C, Tan KBC, Shukla P, Gardiner PV, Small D, Zhang SD, Gibson DS. Assessment of a dried blood spot C-reactive protein method to identify disease flares in rheumatoid arthritis patients. Sci Rep. 2020 Dec 3;10(1):21089. doi: 10.1038/s41598-020-77826-0. PMID 33273485